CLINICAL TRIAL: NCT07360899
Title: Left Atrial Appendage Closure During Cardiac Surgery in Atrial Fibrillation Patients With Seralene
Brief Title: Atrial Fibrillation TRIal of Left Atrial Appendage Closure Using Seralene Hemostatic Suture
Acronym: ATRI-LASH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Cardiovascular Diseases, Vojvodina (Other)
Collaborators: Institute for Cardiovascular Diseases Dedinje (Other); KBC Rebro Zagreb (Unknown); Clinical Centre of Serbia (Other)
Responsible Party: Principal Investigator, Lazar Velicki, Professor, Senior Attending Cardiac Surgeon, Institute of Cardiovascular Diseases, Vojvodina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1351-1/7
Record Dates: First submitted 2026-01-06; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: ATRIAL APPENDAGE CLOSURE for ATRIAL FIBRILLATION; Atrial Fibrillation (AF); Mitral Valve Surgery; Stroke (in Patients With Atrial Fibrillation); Anticoagulant Therapy
MeSH Terms: conditions — Atrial Fibrillation; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AF patients submitted to cardiac surgery (Experimental): Participants in this arm are patients with atrial fibrillation undergoing cardiac surgery for a clinical indication and with a CHA₂DS₂-VASc score of 2 or greater. During the planned cardiac surgical procedure, surgical closure of the left atrial appendage is performed using the CE-marked AtriLASH suture-based device. The intervention is carried out as part of the same operative session and in addition to the indicated cardiac surgery. All participants receive the same intervention.
  Interventions: Device: LAA closure using the AtriLASH

INTERVENTIONS:
Device: LAA closure using the AtriLASH — The intervention consists of surgical closure of the left atrial appendage using the AtriLASH device during cardiac surgery. AtriLASH is a CE-marked, suture-based medical device made of Seralene material and is designed for epicardial closure of the left atrial appendage.
  The device is applied intraoperatively as part of the planned cardiac surgical procedure in patients with atrial fibrillation. The left atrial appendage is identified and closed using the AtriLASH system according to the manufacturer's instructions for use. No additional incisions or separate procedures are required beyond those necessary for the indicated cardiac surgery.
  The intervention is performed in all participants allocated to the study arm and is intended to achieve complete exclusion of the left atrial appendage to reduce the potential for blood stasis and thrombus formation.

SUMMARY:
Atrial fibrillation is a common heart rhythm disorder that increases the risk of stroke. In patients with atrial fibrillation, blood clots most often form in a small structure of the heart called the left atrial appendage. If a blood clot travels from the heart to the brain, it can cause a stroke.

Blood-thinning medications are commonly prescribed to reduce the risk of stroke in patients with atrial fibrillation. However, some patients cannot take these medications long-term because of bleeding risk, side effects, or other medical reasons.

Closing the left atrial appendage is an alternative approach to reduce the risk of stroke by preventing blood from collecting in this area. When patients undergo cardiac surgery for another indication, closure of the left atrial appendage can be performed during the same operation.

This study is designed to evaluate the safety and effectiveness of surgical closure of the left atrial appendage using a device called AtriLASH during cardiac surgery. AtriLASH is a surgical suture-based device intended to close the left atrial appendage.

The study will assess whether the left atrial appendage can be safely and effectively closed using this method in patients with atrial fibrillation undergoing cardiac surgery. The information obtained from this study may help determine whether this approach can reduce the risk of stroke and potentially decrease the need for long-term use of blood-thinning medications in selected patients.

ELIGIBILITY:
Inclusion Criteria:

Age 18 years or older

Documented atrial fibrillation (any type)

CHA₂DS₂-VASc score of 2 or greater, or equivalent stroke risk

Scheduled to undergo cardiac surgery (including coronary artery bypass grafting, valve surgery, or other structural cardiac surgery)

Ability to understand the study and provide written informed consent

Exclusion Criteria:

Contraindication to left atrial appendage closure (e.g., presence of left atrial appendage thrombus or unsuitable anatomy)

Life expectancy less than 3 months, based on clinical judgment

Current participation in another clinical study that could interfere with the outcomes of this study

Active or suspected infective endocarditis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Left atrial appendage patency rate following closure | Three months after the LAA closure
  To evaluate the patency rate of the left atrial appendage (LAA) following closure during cardiac surgery at the 3-month follow-up.

SECONDARY OUTCOMES:
Composite incidence of stroke, systemic embolism, major bleeding, and all-cause mortality | Three months post-surgery
  To assess the safety and efficacy of LAA closure during cardiac surgery in terms of: (1) Incidence of stroke or systemic embolism within 3 months post-surgery.
  (2) Major bleeding events within 3 months post-surgery. (3) All-cause mortality within 3 months post-surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of cardiovascular diseases Vojvodina, Kamenitz, Vojvodina, Serbia

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, ICF, CSR

REFERENCES:
- [Background] Joglar JA, Chung MK, Armbruster AL, Benjamin EJ, Chyou JY, Cronin EM, Deswal A, Eckhardt LL, Goldberger ZD, Gopinathannair R, Gorenek B, Hess PL, Hlatky M, Hogan G, Ibeh C, Indik JH, Kido K, Kusumoto F, Link MS, Linta KT, Marcus GM, McCarthy PM, Patel N, Patton KK, Perez MV, Piccini JP, Russo AM, Sanders P, Streur MM, Thomas KL, Times S, Tisdale JE, Valente AM, Van Wagoner DR; Peer Review Committee Members. 2023 ACC/AHA/ACCP/HRS Guideline for the Diagnosis and Management of Atrial Fibrillation: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2024 Jan 2;149(1):e1-e156. doi: 10.1161/CIR.0000000000001193. Epub 2023 Nov 30. PMID 38033089
- [Background] Tzikas A, Holmes DR Jr, Gafoor S, Ruiz CE, Blomstrom-Lundqvist C, Diener HC, Cappato R, Kar S, Lee RJ, Byrne RA, Ibrahim R, Lakkireddy D, Soliman OI, Nabauer M, Schneider S, Brachmann J, Saver JL, Tiemann K, Sievert H, Camm AJ, Lewalter T. Percutaneous left atrial appendage occlusion: the Munich consensus document on definitions, endpoints, and data collection requirements for clinical studies. Europace. 2017 Jan;19(1):4-15. doi: 10.1093/europace/euw141. Epub 2016 Aug 18. PMID 27540038
- [Background] De Caterina R, Camm AJ. What is 'valvular' atrial fibrillation? A reappraisal. Eur Heart J. 2014 Dec 14;35(47):3328-35. doi: 10.1093/eurheartj/ehu352. Epub 2014 Sep 28. No abstract available. PMID 25265975
- [Background] Ostermayer SH, Reisman M, Kramer PH, Matthews RV, Gray WA, Block PC, Omran H, Bartorelli AL, Della Bella P, Di Mario C, Pappone C, Casale PN, Moses JW, Poppas A, Williams DO, Meier B, Skanes A, Teirstein PS, Lesh MD, Nakai T, Bayard Y, Billinger K, Trepels T, Krumsdorf U, Sievert H. Percutaneous left atrial appendage transcatheter occlusion (PLAATO system) to prevent stroke in high-risk patients with non-rheumatic atrial fibrillation: results from the international multi-center feasibility trials. J Am Coll Cardiol. 2005 Jul 5;46(1):9-14. doi: 10.1016/j.jacc.2005.03.042. PMID 15992628
- [Background] Massumi A, Chelu MG, Nazeri A, May SA, Afshar-Kharaghan H, Saeed M, Razavi M, Rasekh A. Initial experience with a novel percutaneous left atrial appendage exclusion device in patients with atrial fibrillation, increased stroke risk, and contraindications to anticoagulation. Am J Cardiol. 2013 Mar 15;111(6):869-73. doi: 10.1016/j.amjcard.2012.11.061. Epub 2013 Jan 9. PMID 23312129
- [Background] Boersma LV, Schmidt B, Betts TR, Sievert H, Tamburino C, Teiger E, Pokushalov E, Kische S, Schmitz T, Stein KM, Bergmann MW; EWOLUTION investigators. Implant success and safety of left atrial appendage closure with the WATCHMAN device: peri-procedural outcomes from the EWOLUTION registry. Eur Heart J. 2016 Aug;37(31):2465-74. doi: 10.1093/eurheartj/ehv730. Epub 2016 Jan 27. PMID 26822918
- [Background] Holmes DR Jr, Kar S, Price MJ, Whisenant B, Sievert H, Doshi SK, Huber K, Reddy VY. Prospective randomized evaluation of the Watchman Left Atrial Appendage Closure device in patients with atrial fibrillation versus long-term warfarin therapy: the PREVAIL trial. J Am Coll Cardiol. 2014 Jul 8;64(1):1-12. doi: 10.1016/j.jacc.2014.04.029. PMID 24998121
- [Background] Reddy VY, Doshi SK, Sievert H, Buchbinder M, Neuzil P, Huber K, Halperin JL, Holmes D; PROTECT AF Investigators. Percutaneous left atrial appendage closure for stroke prophylaxis in patients with atrial fibrillation: 2.3-Year Follow-up of the PROTECT AF (Watchman Left Atrial Appendage System for Embolic Protection in Patients with Atrial Fibrillation) Trial. Circulation. 2013 Feb 12;127(6):720-9. doi: 10.1161/CIRCULATIONAHA.112.114389. Epub 2013 Jan 16. PMID 23325525
- [Background] Whitlock RP, Vincent J, Blackall MH, Hirsh J, Fremes S, Novick R, Devereaux PJ, Teoh K, Lamy A, Connolly SJ, Yusuf S, Carrier M, Healey JS. Left Atrial Appendage Occlusion Study II (LAAOS II). Can J Cardiol. 2013 Nov;29(11):1443-7. doi: 10.1016/j.cjca.2013.06.015. Epub 2013 Sep 20. PMID 24054920

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-07-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT07360899/Prot_SAP_000.pdf
  • Informed Consent Form (2025-10-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT07360899/ICF_001.pdf